CLINICAL TRIAL: NCT06091267
Title: An Open-label, Crossover, Pharmacokinetic and Efficacy Bridging Study of Oral ASTX727 Versus IV Decitabine in Chinese Subjects With Myelodysplastic Syndromes
Brief Title: PK/Efficacy Bridging Study of ASTX727 in Chinese Subjects With Myelodysplastic Syndromes
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 393-403-00072
Record Dates: First submitted 2023-09-22; First posted 2023-10-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine; decitabine and cedazuridine drug combination; cedazuridine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ASTX727 and IV Decitabine (Experimental): Cycle1：ASTX727 tablets, oral, 1 tablet/day for 5 days；Cycle2：IV Decitabine, 20 mg/m^2, is administered for 1 hour at a time for 5 days；≥ Cycle 3：ASTX727 tablets, oral, 1 tablet/day for 5 days
  Interventions: Drug: IV Decitabine; Drug: Decitabine and cedazuridine; Drug: only Decitabine and cedazuridine
- IV Decitabine and ASTX727 (Active Comparator): Cycle1：IV Decitabine, 20 mg/m^2, is administered for 1 hour at a time for 5 days； Cycle2：ASTX727 tablets, oral, 1 tablet/day for 5 days；≥ Cycle 3：ASTX727 tablets, oral, 1 tablet/day for 5 days
  Interventions: Drug: IV Decitabine; Drug: Decitabine and cedazuridine; Drug: only Decitabine and cedazuridine
- ASTX727 (Experimental): ASTX727 tablets, oral, 1 tablet/day for 5 days；
  Interventions: Drug: only Decitabine and cedazuridine

INTERVENTIONS:
Drug: IV Decitabine — The subjects will receive decitabine 20 mg/m^2 IV daily × 5 days in 28-day cycles.
  Arms: ASTX727 and IV Decitabine; IV Decitabine and ASTX727
Drug: Decitabine and cedazuridine — subjects will receive treatment with ASTX727, 1 tablet/day for 5 consecutive days, in 28-day cycles.
  Arms: ASTX727 and IV Decitabine; IV Decitabine and ASTX727
Drug: only Decitabine and cedazuridine — subjects will receive treatment with ASTX727, 1 tablet/day for 5 consecutive days, in 28-day cycles, until disease progression, unacceptable toxicity, or the subject/investigator decides that the subject should discontinue treatment or withdraw from the trial.

SUMMARY:
This is an Open-Label, Crossover, Pharmacokinetic and Efficacy Bridging Study of Oral ASTX727 versus IV Decitabine in Chinese Subjects with Myelodysplastic Syndromes

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate in this trial and voluntarily sign the informed consent form.
2. Men or women ≥ 18 years at the time of signing the informed consent form.
3. Subjects with MDS previously treated or untreated with de novo or secondary MDS.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at screening.

Exclusion Criteria:

1. Prior treatment with more than 1 cycle of azacitidine or decitabine.
2. Cytotoxic chemotherapy or prior azacitidine or decitabine within 4 weeks of first dose of study treatment.
3. Conditions as judged by the investigator to be inappropriate for participation in the clinical trial.
4. Previous diagnosis of malignant tumor.
5. History of immune deficiency.
6. Acute myeloid leukemia (AML) with bone marrow or peripheral blast count ≥ 20% or other malignant hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | An analysis is planned when the last enrolled patient have completed Follow-up 12 months.
  Assess efficacy [Complete Response Rate (CR)] of treatment with ASTX727 in Chinese subjects with myelodysplastic syndromes (MDS);
5day_AUC0-τ | An analysis is planned when the last enrolled patient have completed the treatment with ASTX727 (oral) versus decitabine for IV infusion for 5 day.
  Assess pharmacokinetic (PK) parameters (Total 5-day AUC exposures of decitabine) after treatment with ASTX727 (oral) versus decitabine for IV infusion for 5 days;

SECONDARY OUTCOMES:
Objective Response Rate | through study completion, an average of 1 year.
  Objective Response Rate (ORR): The proportion of subjects who achieve CR and partial response (PR) based on IWG 2006 criteria;
Clinical Response Rate | through study completion, an average of 1 year.
  Clinical Response Rate: The proportion of subjects who achieve CR, PR, marrow complete response (mCR), and hematologic improvement (HI) based on IWG 2006 criteria.
Rate of transfusion independence | through study completion, an average of 1 year.
  Rate of transfusion independence: The proportion of subjects who had no blood transfusion of 2 or more units of PRBCs for 56 days or more after treatment;
disease progression | through study completion, an average of 1 year.
  Time to progression to acute myeloid leukemia (AML);
Overall survival | through study completion, an average of 1 year.
  Overall survival (OS).
Safety assessment | through study completion, an average of 1 year.
  Safety as assessed by adverse events (AEs), concomitant medications, physical examination, clinical laboratory tests (hematology , serum chemistry and urinalysis), vital signs, Eastern Cooperative Oncology Group (ECOG) performance status, and electrocardiogram (ECG).
peak concentration (Cmax) | through study completion, an average of 1 year.
  Decitabine PK parameters: peak concentration (Cmax).
time to peak concentration (Tmax) | through study completion, an average of 1 year.
  Decitabine PK parameters: time to peak concentration (Tmax).
area under the plasma concentration-time curve over a dosing interval (AUC0-τ). | through study completion, an average of 1 year.
  Decitabine PK parameters: area under the plasma concentration-time curve over a dosing interval (AUC0-τ).
accumulation ratio based on AUC0-τ (Rac_AUC0-τ). | through study completion, an average of 1 year.
  Decitabine PK parameters: accumulation ratio based on AUC0-τ (Rac_AUC0-τ).
accumulation ratio based on Cmax (Rac_Cmax). | through study completion, an average of 1 year.
  Decitabine PK parameters: accumulation ratio based on Cmax (Rac_Cmax).
Cmax | through study completion, an average of 1 year.
  PK parameters of E7727 and E7727-epimer: Cmax.
Tmax | through study completion, an average of 1 year.
  PK parameters of E7727 and E7727-epimer: Tmax.
AUC0-τ | through study completion, an average of 1 year.
  PK parameters of E7727 and E7727-epimer: area under the plasma concentration-time curve over a dosing interval .
Rac_AUC0-τ | through study completion, an average of 1 year.
  PK parameters of E7727 and E7727-epimer: accumulation ratio based on AUC0-τ.
Rac_Cmax | through study completion, an average of 1 year.
  PK parameters of E7727 and E7727-epimer: accumulation ratio based on Cmax.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang, China